CLINICAL TRIAL: NCT05335265
Title: Is Virtual Inhaler Training Successful in COPD?
Brief Title: A Comparison of Classic and Virtual Inhaler Training Methods in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Baha (Other)
Responsible Party: Sponsor-Investigator, Ayse Baha, Associate Professor, MD, Near East University, Turkey
Organization: Near East University, Turkey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YDU/2021/89-1302
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: COPD; Inhaler Training; Face-to-face Training; Video-mediated Virtual Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients randomized according to a simple random numbers table, half of the patients received video-mediated virtual inhaler training (which is published on the Turkish Thoracic Society's official site and with permission for use obtained) and the other half received classical face-to-face inhaler training.
  "Envelope" method was used in randomization.
  -Each clinic prepared 12 envelopes, 6 of them have a paper with the words VIRTUAL EDUCATION and 6 of them CLASSIC EDUCATION. The patient was asked to draw one of these mixed envelopes. The form of education in the envelope was applied to the patient.
Masking Description: "Envelope" method was used in randomization.
  -Each clinic prepared 12 envelopes, 6 of them have a paper with the words VIRTUAL EDUCATION and 6 of them CLASSIC EDUCATION. The patient was asked to draw one of these mixed envelopes. The form of education in the envelope was applied to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIT (face-to-face inhaler training) (Active Comparator): Face-to-face inhaler training.
  o The trainers watched the Turkish Thoracic Society (TTS) MDI training video before giving the training.
  Training given 3 times on the first day, 2 times on the 2nd day, and once on the 3rd day.
  During discharge, inhaler technic was checked according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared by TTS.
  The trainer and the inhaler technical controller are different.
  Interventions: Other: Treatment training
- VIT (virtual inhaler training) (Experimental): Virtual Training was gave 3 times on the first day, 2 times on the 2nd day, and once on the 3rd day (discharge) by the TTS Virtual training video.
  During discharge, inhaler technics of the patient's were controlled according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared by the TTS.
  o The inhaler technique controller and the trainer are different.
  Interventions: Other: Treatment training

INTERVENTIONS:
Other: Treatment training — Face-to-face:Metered-DoseInhalerTraining gave 3 times on the 1st day, 2 times on the 2nd day, once on the 3rd day.During discharge, inhaler technical evaluation were done according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared by using the Patient's Booklet of the Turkish Thoracic Society (TTS).The people who is evaluate the patient's inhaler technique (IT) on the day of discharge was someone different from the health personnel who provided the training. In IT control, the patient's performance was evaluated simultaneously by 2 observers.
  Video training:Training gave 3 times on the 1st day, 2 times on the 2nd day,once on the 3rd day.The TTS-Virtual Training Video were used.During discharge,inhaler technical evaluation was done same with face-to-face training.The person who is evaluate the patient's IT was someone different from the training personnel.In IT observation,it was used same method with face-to-face training.

SUMMARY:
According to the World Health Organization data, the third most common cause of death in the world, is COPD , a disease that progresses with exacerbations (1). Exacerbations are the most important cause of morbidity and mortality in COPD (2). It is thought that most exacerbations occur (3,4) because highly effective inhaler treatments are unavailable to prevent and treat respiratory symptoms (5,6). However, using inhaler devices correctly can be difficult (jama7,8). Guidelines recommend evaluating and teaching inhaler use technique (5,6). Unfortunately, these are often not implemented, especially in a hospital setting (9,10). Worldwide, 25 billion dollars are spent annually on inhaler drugs, 5-7 billion dollars of which is estimated to be wasted because of incorrect technique. Beyond this financial cost, incorrect inhaler technique is associated with worse symptom control, lower quality of life and increased acute care costs, (11,12,13). Although these shortcomings are known, appropriate educational interventions are unfortunately not been available.

Additionally , patient's access to health services (especially face-to-face communication with recommended health providers) has been largely prevented due to the restrictions/requirements implemented against the pandemic in 2020,such as social isolation, staying away from public environments, and ensuring good personal and social hygiene.

Considering that inhaler training is done face-to-face by doctors or allied health personnel today, many patients did not receive inhaler drug use training. One of the most realistic solutions that we encountered with this pandemic is telemedicine. The use of internet-mediated training, which is a part of telemedicine, has come to the foreground. In a recently published study on chronic airway diseases (asthma and COPD), it was revealed that video-mediated inhaler training is as successful as classical face-to-face training (14).Our aim is to investigate whether video-mediated virtual inhaler training is successful in patients with COPD.

DETAILED DESCRIPTION:
Our aim is to investigate whether video-mediated virtual inhaler training is successful in patients with COPD

METHOD OF WORKING

Patients hospitalized due to COPD exacerbation and are ready to be discharged from the hospital will be included in this multicenter, prospective, randomized controlled study. Patients will be randomized according to a simple random numbers table, half of the patients will receive video-mediated virtual inhaler training (which is published on the Turkish Thoracic Society's official site and with permission for use obtained) and the other half will receive the same method as classical facial inhaler training videos.

Depending on the medical condition of the patients admitted to the ward, training will be implemented from the 24th hour of their hospitalization until their discharge stage, starting with 3 training sessions for 3 consecutive days. Upon hospital discharge, the technique of inhaler use evaluation will be carried out according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared using the Turkish Thoracic Society Patient's Booklet.

In inhaler technique training observation, inhaler technique control of the patient will be performed simultaneously by 2 observers independently (each observer will have a checklist) to demonstrate inter-observer consistency.

The patients will be called for a control appointment one week after hospital discharge, and their inhaler technique will be recorded once more using the "inhaler technique control form" by the same 2 observers independently.

RANDOMIZATION:

* ENVELOPE method will be used in randomization.
* Each clinic will prepare 12 envelopes, 6 of them will have a paper with the words VIRTUAL EDUCATION and 6 of them CLASSIC EDUCATION. The patient will be asked to draw one of these mixed envelopes. The form of education in the envelope will be applied to the patient.

Protocol:

* Before discharge, the patient should receive a Metered-Dose Inhaler (MDI) training for 3 consecutive days.
* Classical education (face-to-face education):

  * The person who will provide this training must be a health worker who is an expert in their field.
  * The health personnel who will provide the training should watch the Turkish Thoracic Society MDI training video before giving the training and convey the steps there to the patient (to ensure the patients receive training on an equal basis with the patient who will receive video training).
  * Training should be given 3 times on the first day, 2 times on the 2nd day, and once on the 3rd day.
  * During discharge, inhaler technical evaluation should be done according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared by using the Patient's Booklet of the Turkish Thoracic Society.
  * The people who will evaluate the patient's inhaler technique on the day of discharge should be someone different from the health personnel who provided the training.
  * In inhaler technique observation, the patient's inhaler technique control should be performed simultaneously by 2 observers independently (each observer will have a checklist) to demonstrate inter-observer consistency.

Virtual training (video training):

* On the first day's training, the video should be watched 3 times a day, on the 2nd day the video should be watched 2 times during the day, on the 3rd day (discharge) the video should be watched once.
* In video training, the Turkish Thoracic Society Virtual Training Video, (a copy of the video has been provided ), will be used.
* During discharge, inhaler technical evaluation should be done according to the "Application Steps of Inhalation Techniques Evaluation Form checklist" prepared by using the Patient's Booklet of the Turkish Thoracic Society.
* The people who will evaluate the patient's inhaler technique on the day of discharge should be someone different from the health personnel who provided the training.
* In inhaler technique observation, the patient's inhaler technique control should be performed simultaneously by 2 observers independently (each observer will have a checklist) to demonstrate inter-observer consistency.

  * Upon hospital discharge, the patient should be prescribed a short-acting bronchodilator MDI (This is already recommended for all patients in Groups A, B, C, and D according to the GOLD guidelines. In this respect, our study does not fall under a drug study).
  * They should not be advised to watch or not watch the Inhaler Training Video at home (If we allow them to access and watch the video at home, it will create bias). The decision of whether to watch the video at home should be left to the patient (a question will be asked about this at the control. It has been added to the form).
  * The first control after discharge should be done in the 1st week. Patients who cannot come to the hospital for a control appointment due to the pandemic will be called by phone and inhaler techniques will be checked with video conversation. (There is no legal issues as no image recording will be taken here).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not used MDI for at least 1 year.
* Having COPD diagnosed with PFT (FEV1/FVC <70 in PFT in the last 1 year)
* Being hospitalized with a COPD exacerbation and being discharged
* Not having a hearing loss, mental disability, visual impairment and a physical impairment that would prevent the use of MDI
* To have the necessary technological equipment to establish video communication on the phone
* Who have agreed to participate in the study.

Exclusion Criteria:

* Patients who have used MDI or have training MDI for at least 1 year.
* Having a hearing loss, mental disability, visual impairment and a physical impairment that would prevent the use of MDI
* Have not the necessary technological equipment to establish video communication on the phone

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The success of virtual education | 2 weeks
  The primary outcome is to investigate whether video-mediated virtual inhaler training is successful in patients with COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Ayse Baha, Study Chair — Near East University Faculty of Medicine; Dilek Yapar, Principal Investigator — Antalya Muratpasa District Health Directorate; Aylin O Alpaydin, Principal Investigator — Dokuz Eylül University Faculty of Medicine; Aycan Yuksel, Principal Investigator — Ufuk University; Ayshan Mammadova, Principal Investigator — Gazi University Faculty of Medicine; Ali Uzan, Principal Investigator — Near East University Faculty of Medicine; Deniz Kizilirmak, Principal Investigator — Celal Bayar University Faculty of Medicine; Esen S Gulensoy, Principal Investigator — Ufuk University; İlknur Kaya, Principal Investigator — Kütahya Faculty of Health Science; Irem Serifoglu, Principal Investigator — Ankara City Hospital Bilkent; Ismail Zehir, Principal Investigator — Kütahya Faculty of Science; Merve Y Senel, Principal Investigator — Balıkesir State Hospital; Nalan Ogan, Principal Investigator — Ufuk University; Nurdan Kokturk, Principal Investigator — Gazi University Faculty of Medicine; Secil Sari, Principal Investigator — Celal Bayar University Faculty of Medicine; Umran O Sertcelik, Principal Investigator — Ankara City Hospiatl; Zuleyha Galata, Principal Investigator — Gazi University Faculty of Medicine
Locations (9):
- Turkey (Türkiye) (9):
  - Ankara City Hospital, Ankara
  - Gazi University Faculty of Medicine, Ankara
  - Ufuk University Faculty of Medicine, Ankara
  - Muratpasa District Health Directorate, Antalya
  - Balıkesir State Hospital, Balıkesir
  - Dokuz Eylul University, Faculty of Medicine, Izmir
  - Kütahya University of Health Sciences, Kütahya
  - Celal Bayar University Faculty of Medicine, Manisa
  - Near East University Faculty of Medicine, Mersin-10

IPD SHARING:
Plan to Share IPD: No